CLINICAL TRIAL: NCT05660759
Title: N-butyl-cyanoacrylate Glue Versus Micro Particles and the Effect on Inducing Liver Hypertrophy After Portal Vein Embolization- a Retrospective Swedish Multicenter Study
Brief Title: Comparison of N-butyl-cyanoacrylate and Micro Parti-cles Effect in Inducing Liver Hypertrophy After PVE
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Karolinska Institutet (Other); Skane University Hospital (Other)
Responsible Party: Principal Investigator, Bergthor Björnsson, Professor, Linkoeping University
Other Study IDs: DB_01
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Portal Vein Embolization, Liver, Hypertrophy
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NBCA: Patients that recieved portal vein embolization with n-butyl-cyanoacrylate glue.
  Interventions: Procedure: Portal vein embolization
- Particles: Patients that recieved portal vein embolization with micro particles.
  Interventions: Procedure: Portal vein embolization

INTERVENTIONS:
Procedure: Portal vein embolization — Portal vein emboliazation with either NBCA or micro particles.

SUMMARY:
The aim of this study is to compare hypertrophy of the FLR after PVE with microparticles to hypertrophy after PVE with cyanoacrylate in a material large enough to answer the study question. In addition, other factors that may influence the degree of hypertrophy will be evaluated in a multivariable analysis.

The hypothesis is: PVE with cyanoacrylate is superior to PVE with microparticles in terms of FLR hy-pertrophy.

DETAILED DESCRIPTION:
With expansion of indications for major liver surgery, portal vein embolization (PVE) is increasingly used in order to induce hypertrophy of the future liver remnant (FLR). De-spite vide variety of materials available to occlude the portal veins the most commonly used are cyanoacrylate and microparticles/spheres. Earlier studies have failed to show superiority of one over the other in terms of hypertrophy of the FLR while PVE with cy-anoacrylate seems to be less time consuming. Two small previous studies from single centers have shown greater growth by cyanoacrylate compared to particles (1) with 90 included patients and the second study with 34 included patients (2), but larger reviews have failed (3). Cyanoacrylate might give a more robust FLR hypertrophy (4) . The main problem in evaluating previous studies has been the large heterogeneity and the often poorly described study populations.

ELIGIBILITY:
Inclusion Criteria: Over 18 years old. Planned for portal vein embolization. -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing portal vein embolization during the study period 2013 - 2021 in Linköping University Hospital, Karolinska Comprehensive Cancer Center and Skåne University Hospital Lund.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
FLR hypertrophy | Spring 2023

SECONDARY OUTCOMES:
Degree of hypertrophy | Spring 2023
Kinetic growth rate | Spring 2023

CONTACTS AND LOCATIONS:
Overall Officials: Bergthor Björnsson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided